CLINICAL TRIAL: NCT03001362
Title: Radical External Beam Chemoradiation in Patients With Rectal Cancer: a "Wait-and-see" Approach
Brief Title: Patients With Rectal Cancer: a "Wait-and-see" Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Neil Kopek, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-407 GEN
Record Dates: First submitted 2016-12-14; First posted 2016-12-23 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radical External Beam RT for Colorectal Ca (Experimental): A single arm consisting of: Radical external beam RT dose of 54 Gy in 30fx with radiosensitizing chemotherapy as per institutional standard
  Interventions: Radiation: Radical external beam radiotherapy

INTERVENTIONS:
Radiation: Radical external beam radiotherapy — pelvic radiotherapy to a dose of 45 Gy in 25 fractions with a tumor boost to a dose of 9 Gy in 5 fractions (thus total of 54 Gy/30 fractions to the primary tumor), combined with radio sensitizing chemotherapy.
  Other Names: Radiosensitizing chemotherapy

SUMMARY:
Patients with histologically proven adenocarcinoma of the rectum will receive pelvic radiotherapy to a dose of 45Gy in 25 fractions with a tumor boost to a dose of 9Gy in 5 fractions (thus total of 54Gy/30Fx to the primary tumor), combined with radio sensitizing chemotherapy. Patients will then be closely monitored, through endoscopy and imaging, for response to treatment and relapse. Salvage oncologic surgery to be offered if there is failure to achieve complete clinical response or in the event of a loco regional relapse.

DETAILED DESCRIPTION:
The combination of preoperative (chemo)radiotherapy and total mesorectal excision (TME) has been shown to reduce the risk of local recurrence in patients with resectable adenocarcinoma of the rectum. The improved local control rates come at the price of an increased risk of surgical complications, including a postoperative death rate of 2-8 percent which may reach 30 per cent at 6 months in those aged over 85 years, as well as long-term impact on anorectal, urinary and sexual function. Patients with cancers in the low rectum in close proximity to the sphincter muscles, may require a permanent stoma, which can be associated with high psychological morbidity.

Preoperative chemoradiotherapy followed by a delay to resection can produce pathological complete responses. One review of phase II and III studies identified an overall pCR rate of 13.5%, but even higher rates of pCR have been observed with doses of radiotherapy exceeding 45 Gy . Certainly patients who proceed to radical surgery after achieving a pCR with chemo radiation do have favorable long-term outcomes. But do patients whose tumor has already been sterilized by chemo radiotherapy need to proceed with radical surgery?

A number of studies have now emerged highlighting the rationale of a 'wait and see' policy for patients who achieve a complete clinical response (cCR) after chemo radiotherapy. The majority of the clinical data supporting this approach have come from Brazil. The Brazilian data suggests that observation of such patients yields survival rates similar to those of patients who undergo radical surgery with confirmation of pCR. More recent studies from the United Kingdom and the Netherlands appear to support the feasibility of this approach. To date there is no published prospectively collected data of a wait-and-see policy from a North American Centre.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic MRI defined disease (at least one of the following):

  * mesorectum involved or breached - includes involvement of adjacent organ (s) (T3-T4)
  * involvement of muscularis propria (T2)
  * extra-mural vascular invasion
  * tumour deposit within the mesorectum
  * one or more involved mesorectal lymph node
* Patients are considered medically fit for oncologic resection
* ECOG performance status 0 or 1
* No evidence of established metastatic disease (CT chest and abdomen)
* Absolute neutrophil count >1.5x109/L; platelets >100x109/L,
* Serum transaminase <3 x ULN;
* Adequate renal function (Cockroft Gault estimation >50 mL/min)
* Bilirubin <1.5 x ULN
* Ability to comply with oral medication
* Willingness and ability to give informed consent and comply with treatment and follow up schedule
* Age 18 or over

Exclusion Criteria:

* Previous radiotherapy to the pelvis (including brachytherapy)
* Enlarged extramesorectal nodes
* Uncontrolled cardiorespiratory comorbidity (includes patients with inadequately controlled angina or myocardial infarction within 6 months of randomisation)
* T1N0 disease without extra-mural venous invasion
* Unequivocal evidence of metastatic disease (includes resectable metastases)
* Major impairment of bowel function without defunctioning stoma/ileostomy (baseline grade 3 diarrhoea or clinically significant faecal incontinence)
* History of another malignancy within the last 5 years except successfully treated basal cell cancer of skin or carcinoma in situ of uterine cervix.
* Known dihydropyrimidine dehydrogenase deficiency
* Known Gilberts disease (hyperbilirubinaemia)
* Taking warfarin or phenytoin or sorivudine
* Gastrointestinal disorder which would interfere with oral therapy and its bioavailability
* Pregnant, lactating, or pre-menopausal women not using adequate contraception
* Unfit to receive any study treatment or subsequent surgical resection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a "wait and see" approach | One year
  Rate of failure to achieve CR or the rate of recurrence after achieving CR

CONTACTS AND LOCATIONS:
Overall Officials: Neil Kopek, M.D., Principal Investigator — Radiation Oncologist
Locations (2):
- Canada (2):
  - McGill University Health Center-Cedars Cancer Centre, Montreal, Quebec
  - McGill University Health Centre- Cedars Cancer Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Background] Peeters KC, Marijnen CA, Nagtegaal ID, Kranenbarg EK, Putter H, Wiggers T, Rutten H, Pahlman L, Glimelius B, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. The TME trial after a median follow-up of 6 years: increased local control but no survival benefit in irradiated patients with resectable rectal carcinoma. Ann Surg. 2007 Nov;246(5):693-701. doi: 10.1097/01.sla.0000257358.56863.ce. PMID 17968156
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Borowski DW, Bradburn DM, Mills SJ, Bharathan B, Wilson RG, Ratcliffe AA, Kelly SB; Northern Region Colorectal Cancer Audit Group (NORCCAG). Volume-outcome analysis of colorectal cancer-related outcomes. Br J Surg. 2010 Sep;97(9):1416-30. doi: 10.1002/bjs.7111. PMID 20632311
- [Background] Paun BC, Cassie S, MacLean AR, Dixon E, Buie WD. Postoperative complications following surgery for rectal cancer. Ann Surg. 2010 May;251(5):807-18. doi: 10.1097/SLA.0b013e3181dae4ed. PMID 20395841
- [Background] Rutten HJ, den Dulk M, Lemmens VE, van de Velde CJ, Marijnen CA. Controversies of total mesorectal excision for rectal cancer in elderly patients. Lancet Oncol. 2008 May;9(5):494-501. doi: 10.1016/S1470-2045(08)70129-3. PMID 18452860
- [Background] Bujko K, Nowacki MP, Nasierowska-Guttmejer A, Michalski W, Bebenek M, Kryj M. Long-term results of a randomized trial comparing preoperative short-course radiotherapy with preoperative conventionally fractionated chemoradiation for rectal cancer. Br J Surg. 2006 Oct;93(10):1215-23. doi: 10.1002/bjs.5506. PMID 16983741
- [Background] Gervaz PA, Wexner SD, Pemberton JH. Pelvic radiation and anorectal function: introducing the concept of sphincter-preserving radiation therapy. J Am Coll Surg. 2002 Sep;195(3):387-94. doi: 10.1016/s1072-7515(02)01308-x. No abstract available. PMID 12229948
- [Background] Hartley A, Ho KF, McConkey C, Geh JI. Pathological complete response following pre-operative chemoradiotherapy in rectal cancer: analysis of phase II/III trials. Br J Radiol. 2005 Oct;78(934):934-8. doi: 10.1259/bjr/86650067. PMID 16177017
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Habr-Gama A, Perez RO, Proscurshim I, Campos FG, Nadalin W, Kiss D, Gama-Rodrigues J. Patterns of failure and survival for nonoperative treatment of stage c0 distal rectal cancer following neoadjuvant chemoradiation therapy. J Gastrointest Surg. 2006 Dec;10(10):1319-28; discussion 1328-9. doi: 10.1016/j.gassur.2006.09.005. PMID 17175450
- [Background] Habr-Gama A, Perez RO, Nadalin W, Sabbaga J, Ribeiro U Jr, Silva e Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Operative versus nonoperative treatment for stage 0 distal rectal cancer following chemoradiation therapy: long-term results. Ann Surg. 2004 Oct;240(4):711-7; discussion 717-8. doi: 10.1097/01.sla.0000141194.27992.32. PMID 15383798
- [Background] Habr-Gama A, Perez RO, Nadalin W, Nahas SC, Ribeiro U Jr, Silva E Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Long-term results of preoperative chemoradiation for distal rectal cancer correlation between final stage and survival. J Gastrointest Surg. 2005 Jan;9(1):90-9; discussion 99-101. doi: 10.1016/j.gassur.2004.10.010. PMID 15623449
- [Background] Habr-Gama A, Gama-Rodrigues J, Sao Juliao GP, Proscurshim I, Sabbagh C, Lynn PB, Perez RO. Local recurrence after complete clinical response and watch and wait in rectal cancer after neoadjuvant chemoradiation: impact of salvage therapy on local disease control. Int J Radiat Oncol Biol Phys. 2014 Mar 15;88(4):822-8. doi: 10.1016/j.ijrobp.2013.12.012. Epub 2014 Feb 1. PMID 24495589
- [Background] Habr-Gama A, de Souza PM, Ribeiro U Jr, Nadalin W, Gansl R, Sousa AH Jr, Campos FG, Gama-Rodrigues J. Low rectal cancer: impact of radiation and chemotherapy on surgical treatment. Dis Colon Rectum. 1998 Sep;41(9):1087-96. doi: 10.1007/BF02239429. PMID 9749491
- [Background] Habr-Gama A. Assessment and management of the complete clinical response of rectal cancer to chemoradiotherapy. Colorectal Dis. 2006 Sep;8 Suppl 3:21-4. doi: 10.1111/j.1463-1318.2006.01066.x. PMID 16813588
- [Background] Dalton RS, Velineni R, Osborne ME, Thomas R, Harries S, Gee AS, Daniels IR. A single-centre experience of chemoradiotherapy for rectal cancer: is there potential for nonoperative management? Colorectal Dis. 2012 May;14(5):567-71. doi: 10.1111/j.1463-1318.2011.02752.x. PMID 21831177
- [Background] Maas M, Beets-Tan RG, Lambregts DM, Lammering G, Nelemans PJ, Engelen SM, van Dam RM, Jansen RL, Sosef M, Leijtens JW, Hulsewe KW, Buijsen J, Beets GL. Wait-and-see policy for clinical complete responders after chemoradiation for rectal cancer. J Clin Oncol. 2011 Dec 10;29(35):4633-40. doi: 10.1200/JCO.2011.37.7176. Epub 2011 Nov 7. PMID 22067400
- [Background] Glynne-Jones R, Hughes R. Critical appraisal of the 'wait and see' approach in rectal cancer for clinical complete responders after chemoradiation. Br J Surg. 2012 Jul;99(7):897-909. doi: 10.1002/bjs.8732. Epub 2012 Apr 27. PMID 22539154
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Temple LK, Bacik J, Savatta SG, Gottesman L, Paty PB, Weiser MR, Guillem JG, Minsky BD, Kalman M, Thaler HT, Schrag D, Wong WD. The development of a validated instrument to evaluate bowel function after sphincter-preserving surgery for rectal cancer. Dis Colon Rectum. 2005 Jul;48(7):1353-65. doi: 10.1007/s10350-004-0942-z. PMID 15868235